CLINICAL TRIAL: NCT03299036
Title: Hydrophilic Radiopaque Microsphere With Doxorubicin for Hepatoma Embolization Therapy
Brief Title: Drug-loadable（T-ACE Beads）for Hepatoma Embolization Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: The Industrial Technology Research Institute (Other); National Cheng Kung University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B-BR-105-054
Record Dates: First submitted 2017-09-20; First posted 2017-10-02 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Cancer of Liver
Keywords: Hepatoma; Transcatheter Arterial chemo-embolization; Microsphere; Doxorubicin
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Taiwan ACE Beads with doxorubicin (Experimental): The use of Taiwan ACE Beads (T-ACE) microspheres embolization with doxorubicin as a treatment for patients with hepatoma.
  Interventions: Device: Taiwan ACE Beads with doxorubicin

INTERVENTIONS:
Device: Taiwan ACE Beads with doxorubicin — Similar with commercializing drug-eluting beads, radiologist inject Taiwan ACE Beads with doxorubicin instead of Gelfoam or polyvinyl alcohol.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Radiopaque Microsphere (T-ACE Beads with doxorubicin) interventional therapy for patients with liver cancer

DETAILED DESCRIPTION:
The study will evaluate the safety and tolerability of Taiwan ACE Beads with doxorubicin used for chemoembolization for the treatment of unresectable hepatocellular carcinoma.

The investigators will study the overall response rates of lesions with Taiwan ACE Beads.

The procedure is similar with the other commercializing drug-eluting beads. At the target vessels, radiologists will inject doxorubicin with Taiwan ACE Beads instead of Gelfoam or PVA (polyvinyl alcohol). The end point of injection is also similar with conventional TACE.

Determine the complication rates, progression free survival (PFS) and overall survival (OS) following Taiwan ACE Beads embolization.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria in order to be entered into the study:

A. Both genders of patients age 20 or older.

B. Patients diagnosed of liver cancer (MUST meet at least ONE of the following criteria:)

1. Diagnosed via tumor biopsy by Pathologists, and confirmed by on-service physician.
2. High risk patients (Viral hepatitis B or C or cirrhotics) with typical liver cancer image appeared on more than two radiographic examinations (Ultrasound, MRI, CT scan or Angiography).
3. High risk patients (Viral hepatitis B or C cirrhotics) with evidence of enlarging image of liver cancer via more than two follow-up records.

C. In intermediate stage by BCLC staging, tumor size under 8 centimeters, with liver function at Child-Pugh class ≤ 8, and is either difficult to accept an operation or reluctant to accept any operation.

D. Disease can be treated by transarterial chemoembolization, and can be evaluated by Ultrasound, Magnetic resonance imaging (MRI), or computed tomography (CT).

E. Performance status ECOG 2 or less. Patient has a life expectancy of at least 3 months.

Exclusion Criteria:

If patients meet any of the following criteria they may not be entered into the study:

A. major branch of portal vein has been invaded already; extrahepatic metastasis or the the other malignant tumors.

B. Evidences of decompensation: Total Bilirubin>2, PT prolong>3 seconds, Child-Pugh class>8, refractory ascites, active bleeding, hepatic encephalopathy, and severe infection.

C. Tumor size (diameter) larger than 8 centimeters.

D. Not on dialysis with Creatinine >2.0 mg/dL.

E. Allergic to iodine or other injections.

F. Other main organ failure (Heart, Lung, or Kidney).

G. WBC<3000, or Platelet Count <50,000 mg/dL.

H. Performance status ECOG of 3 or more.

I. Pregnant women and breath feeding women.

J. Patients whose blood vessel are too difficult to do Taiwan ACE Beads procedure.

K. Prominent AV shunt.

L. Severe atherosclerosis.

M. Vasospasm or possible major vascular injury.

N. Arteriovenous shunt patients, diameter larger than the size of microsphere available.

O. Collateral vascular exists and may endanger non-targeted area during arterial chemoembolization.

P. Contraindications for doxorubicin.

Q. Numerous of tumors locate at different lobes, high risk of Hepatic insufficiency.

R. Unwilling to sign a written informed consent form.

S. Allergic to pharmaceutical excipients related to Microspheres.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-10-16 (Actual); Study Completion 2018-10-16 (Actual)

PRIMARY OUTCOMES:
Patients Survival (Safety) | An average of 12 weeks.
  Survival rate will be evaluated since treatment day until the date of death or final observation.
Tumor response in patients with hepatoma who received Taiwan ACE beads (TACE) microspheres embolization evaluated with mRECIST criteria | Three months
  mRECIST criteria will be used to evaluate tumor response in patients with hepatoma who received Taiwan ACE beads (TACE) microspheres embolization.

SECONDARY OUTCOMES:
Serum Level of AFP | An average of 12 weeks
  Collect Doxorubicin's blood concentration, 5 mL each time

CONTACTS AND LOCATIONS:
Overall Officials: Xi-Zhang Lin, Study Director — Department of Internal Medicine, National Cheng Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu YS, Lin XZ, Tsai HM, Tsai HW, Chen GC, Chen SF, Kang JW, Chou CM, Chen CY. Development of biodegradable radiopaque microsphere for arterial embolization-a pig study. World J Radiol. 2015 Aug 28;7(8):212-9. doi: 10.4329/wjr.v7.i8.212. PMID 26339465
- [Background] Liu YS, Ou MC, Tsai YS, Lin XZ, Wang CK, Tsai HM, Chuang MT. Transarterial chemoembolization using gelatin sponges or microspheres plus lipiodol-doxorubicin versus doxorubicin-loaded beads for the treatment of hepatocellular carcinoma. Korean J Radiol. 2015 Jan-Feb;16(1):125-32. doi: 10.3348/kjr.2015.16.1.125. Epub 2015 Jan 9. PMID 25598680